CLINICAL TRIAL: NCT03224819
Title: A Phase 1 First-In-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of AMG 673 Administered as Short Term Intravenous Infusions in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study of Emerfetamab (AMG 673) in Adults With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Priortization of other Programs
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160377; 2017-002980-16 (EudraCT Number)
Record Dates: First submitted 2017-07-03; First posted 2017-07-21 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Bayesian Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): The dose-escalation cohorts to estimate the MTD will use 2 schedules of emerfetamab administration: Schedule A (Day 1/Day 5 dosing in 14-day cycles) and Schedule B (once daily dosing for cycle 1 followed by twice weekly dosing in following cycles).
  For Schedule A the starting dose for the first cohort will be 0.05 μg emerfetamab administered as short term IV infusions on day 1 and day 5. The doses administered for the following cohorts will be recommended by the Dose Level Review Team (DLRT).
  For Schedule B the starting dose will be 72 μg emerfetamab administered as short-term IV infusions daily (QD) during the 14-day cycle 1 after the 72 μg target dose is found to be relatively safe and tolerable by the DLRT for Schedule A.
  Interventions: Drug: Emerfetamab
- Expansion Phase (Experimental): For each schedule, upon completion of the dose escalation cohorts, additional participants may be enrolled to receive emerfetamab at a dose at or below the MTD estimated in the dose escalation cohorts.
  Interventions: Drug: Emerfetamab

INTERVENTIONS:
Drug: Emerfetamab — Administered by intravenous (IV) infusion.
  Other Names: AMG 673

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of emerfetamab in adults with relapsed/refractory acute myeloid leukemia (AML) and to estimate the maximum tolerated dose (MTD) and/or a biologically active dose (eg, recommended phase 2 dose [RP2D]).

DETAILED DESCRIPTION:
This is a first-in-human, open-label, phase 1, sequential dose escalation study. Emerfetamab will be evaluated as a short term intravenous (IV) infusion in adults with relapsed/refractory AML The study will consist of a dose escalation phase and a dose expansion phase. The study was terminated prior to the start of the expansion phase.

ELIGIBILITY:
Inclusion Criteria

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Subjects ≥ 18 years of age at the time of signing consent.
* AML as defined by the World Health Organisation (WHO) Classification persisting or recurring following 1 or more treatment courses except promyelocytic leukemia (APML).

  * More than 5% myeloblasts in bone marrow.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.

Exclusion Criteria

* Known hypersensitivity to immunoglobulins.
* Autologous hematopoietic stem cell transplantation (HSCT) within 6 weeks prior to start of AMG 673 treatment.
* Allogeneic HSCT within 3 months prior to start of AMG 673 treatment.
* Non-manageable graft versus host disease.
* Known positive test for human immunodeficiency virus (HIV).
* Males and females of reproductive potential who are unwilling to practice a highly effective method(s) of birth control while on study through 15 weeks after receiving the last dose of study drug. Acceptable methods of highly effective birth control include sexual abstinence (males, females); vasectomy; bilateral tubal ligation/occlusion; or a condom with spermicide (men) in combination with hormonal birth control or intrauterine device (IUD) (women). Males who are unwilling to abstain from sperm donation while on study through 5 half-lives after receiving the (last [multiple-dose studies]) dose of study drug.
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 15 weeks after receiving the last dose of study drug.
* Females with a positive pregnancy test
* Females planning to become pregnant while on study through 15 weeks after receiving the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Klinikum der Ludwig Maximilians Univeritaet, MÃ¼nchen, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in United States, Australia, and Germany.
Groups:
- Schedule A Cohort 1: 0.05 µg Emerfetamab: Participants received 0.05 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 2: 0.15 µg Emerfetamab: Participants received 0.15 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 3: 0.45 µg Emerfetamab: Participants received 0.45 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 4: 1.5 µg Emerfetamab: Participants received 1.5 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 5: 4.5 µg Emerfetamab: Participants received 4.5 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 6: 7 µg Emerfetamab: Participants received 7 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 7: 9 µg Emerfetamab: Participants received 9 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 8: 18 µg Emerfetamab: Participants received 18 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 9: 36 µg Emerfetamab: Participants received 36 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 10: 72 µg Emerfetamab: Participants received 72 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 11: 110 µg Emerfetamab: Participants received 110 µg emerfetamab intravenously on day 1 and day 5 of each 14-day cycle for up to 12 total treatment cycles.
- Schedule A Cohort 12: 36/72 µg Emerfetamab: Participants received 36 µg emerfetamab intravenously on day 1 and 72 µg emerfetamab on day 5 and thereafter of each 14-day cycle for up to 12 total treatment cycles.
- Schedule B Cohort 1: 72 µg Emerfetamab: Participants received 72 µg emerfetamab intravenously once a day (QD) from days 1 to 14 for the first treatment cycle then on day 1, day 4, day 8, and day 11 of each subsequent 14-day cycle for up to a total of 12 cycles.
- Schedule B Cohort 2: 110 µg Emerfetamab: Participants received 72 µg emerfetamab intravenously on day 1 and day 2 then 110 µg emerfetamab once a day from days 3 to 14 in the first treatment cycle, then 110 µg emerfetamab on day 1, day 4, day 8, and day 11 of each subsequent 14-day cycle for up to a total of 12 cycles.
Period: Overall Study
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Started | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3
Completed | 1 | 0 | 3 | 2 | 2 | 1 | 2 | 1 | 2 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 | 61.0 | 49.3 (16.3) | 69.3 (8.1) | 60.3 (23.9) | 60.7 (18.9) | 73.7 (2.1) | 45.7 (14.6) | 68.8 (11.8) | 71.8 (7.0) | 57.5 (11.6) | 72.0 (5.1) | 61.4 (18.2) | 54.0 (7.5) | 62.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 2 | 3 | 3 | 2 | 3 | 2 | 23
  Male | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 2 | 2 | 3 | 1 | 2 | 2 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5
  Not Hispanic or Latino | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3 | 4 | 2 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black (or African American) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 | 3 | 1 | 3 | 3 | 2 | 4 | 6 | 4 | 3 | 4 | 3 | 41
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: The severity of each adverse event (AE) was graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria, where Grade 1 = mild AE, Grade 2 = moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening and Grade 5 = death due to AE.
  A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From first dose of study drug until the end of study; median (minimum, maximum) duration was 1.22 (0.10, 5.98) months.
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3
Participants
  Any treatment emergent adverse event (TEAE) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3
  TEAE Grade ≥ 2 | 1 | 1 | 3 | 3 | 2 | 3 | 2 | 3 | 4 | 6 | 4 | 4 | 5 | 3
  TEAE Grade ≥ 3 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 3 | 3 | 5 | 4 | 4 | 5 | 3
  TEAE Grade ≥ 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 3 | 4 | 2 | 4 | 2
  Serious adverse events (SAE) | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 2 | 5 | 3 | 4 | 1 | 2
  TEAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  SAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  TEAE leading to interruption of study drug | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 2
  SAE leading to interruption of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Fatal adverse events | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Treatment related TEAEs | 1 | 1 | 1 | 3 | 3 | 1 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: A DLT was defined as any of the events described below occurring in a participant during the DLT window, unless clearly attributable to causes other than emerfetamab:
  * Any treatment-related death;
  * Grade 4 neutropenia persisting at 42 days after the last infusion in treatment cycle 1;
  * Grade 3-5 non-hematologic toxicity not clearly resulting from the underlying leukemia with a few protocol-specified exceptions;
  * Grade 2 or 3 cytokine release syndrome (CRS) meeting any of the criteria listed below:
    * Grade 2 CRS that does not resolve, with or without intervention to Grade 1 within 7 days;
    * Grade 3 CRS that does not resolve, with or without intervention to Grade 2 within 5 days, or grade 1 within 7 days;
    * Grade 3 CRS reported at the initial dose;
    * Two separate grade 3 CRS events;
  * Grade 4 CRS occurring during treatment.
Time Frame: Schedule A: From the start of the first infusion on day 1 until day 14. Schedule B: From the start of the first infusion on day 1 to day 28.
Population: Enrolled participants who received at least 1 dose of study drug who received the minimum cycle 1 doses planned for the respective cohort:
  Schedule A: 2 doses within 14-day window; Schedule B: completed ≥ 70% of the planned target doses within 28-day window.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3 | 3 | 3
Participants
  Any dose-limiting toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Acute kidney injury | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bone pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cytokine release syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lipase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Schedule A: Maximum Observed Concentration (Cmax) of Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of pharmacokinetic (PK) parameters. Concentrations below the lower limit of quantitation (LLOQ; 0.0015 ng/mL) were set to zero before data analysis.
Time Frame: Cycle 1 day 1 at predose and at 1, 6, 24, and 48 hours after the start of infusion, and day 5 at predose and 1, 6, 12, 24, 48, 72, and 312 hours after the start of infusion.
Population: Participants who received at least 1 dose of study drug, had at least 1 PK sample collected, with enough data for calculation of the PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4
ng/mL
  Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3
  Day 1 | 0.00979 | 0.038 | 0.0255 (0.0335) | 0.0463 (0.0436) | 0.347 (0.133) | 1.04 (1.43) | 0.960 (1.10) | 1.12 (1.12) | 2.16 (1.78) | 3.15 (1.90) | 4.65 (1.64) | 1.84 (1.08)
  Day 5: number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 5 | 3 | 4
  Day 5 | 0.011 | 0.027 | 0.0448 (0.00672) | 0.0587 (0.0517) | 0.264 (NA) — Not calculated when N=2 | 0.731 (0.529) | 0.961 (1.30) | 1.23 (0.586) | 2.01 (0.926) | 3.14 (1.80) | 5.07 (2.53) | 3.29 (0.484)

4. Secondary Outcome: Schedule A: Time to Maximum Observed Concentration (Tmax) of Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
Time Frame: as for outcome 3
Population: Participants who received at least 1 dose of study drug, had at least 1 pharmacokinetic (PK) sample collected, with enough data for calculation of the PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4
hours
  Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3
  Day 1 | 0.53 | 0.50 | 0.62 [0.38 to 0.75] | 0.48 [0.0 to 0.75] | 0.5 [0.5 to 2.3] | 0.50 [0.35 to 1.8] | 2.0 [0.48 to 6.0] | 1.0 [0.52 to 1.2] | 1.0 [1.0 to 1.2] | 1.1 [0.92 to 2.1] | 1.1 [1.0 to 1.3] | 0.97 [0.62 to 1.2]
  Day 5: number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 5 | 3 | 4
  Day 5 | 4.08 | 2 | 2.3 [1.9 to 2.3] | 2.1 [2.0 to 2.1] | 1.9 [1.7 to 2.0] | 2.0 [1.9 to 2.0] | 1.1 [1.0 to 24] | 1.1 [1.1 to 1.8] | 1.0 [0.95 to 1.1] | 1.1 [0.98 to 6.1] | 1.0 [0.93 to 1.1] | 1.1 [0.98 to 1.5]

5. Secondary Outcome: Schedule A: Area Under the Concentration-time Curve From Time Zero to 96 Hours Post-dose (AUC0-96) on Day 1 for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The area under the curve (AUC) from time zero to 96 hours postdose was calculated using the linear trapezoidal method.
Time Frame: Cycle 1 day 1 at predose and at 1, 6, 24, 48, and 96 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 2 | 3 | 3 | 3 | 3 | 4 | 5 | 4 | 3
hr*ng/mL | 0.222 | 0.84 | 0.659 (0.664) | 1.03 (NA) — Not calculated when N=2 | 5.37 (1.23) | 12.0 (8.79) | 13.5 (10.4) | 16.5 (13.0) | 22.4 (9.66) | 34.4 (11.7) | 62.4 (10.4) | 18.3 (5.02)

6. Secondary Outcome: Schedule A: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Non-compartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The area under the concentration-time curve from time 0 relative to the start of the IV infusion to the last quantifiable concentration was estimated using the linear trapezoidal method.
Time Frame: Cycle 1 day 5 at predose and 1, 6, 12, 24, 48, 72, and 312 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 5 | 3 | 4
hr*ng/mL | 0.302 | 0.745 | 1.38 (0.406) | 1.01 (0.855) | 5.93 (NA) — Not calculated for N = 2 | 22.7 (24.2) | 14.4 (9.69) | 19.3 (8.95) | 27.1 (12.9) | 35.3 (9.13) | 56.8 (31.3) | 35.7 (7.85)

7. Secondary Outcome: Schedule A: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Non-compartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The area under the concentration-time curve from time 0 relative to the start of the IV infusion to infinity was estimated using the linear trapezoidal method.
Time Frame: Cycle 1 day 5 at predose and 1, 6, 12, 24, 48, 72, and 312 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 0 | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 4 | 5 | 3 | 4
hr*ng/mL |  | 0.784 | 1.56 (0.394) | 1.56 (NA) — Not calculated when N=2 | 6.16 (NA) — Not calculated when N=2 | 23.6 (25.1) | 15.3 (10.8) | 16.3 (NA) — Not calculated when N=2 | 28.6 (13.1) | 36.8 (9.04) | 61.0 (36.5) | 38.3 (10.9)

8. Secondary Outcome: Schedule A: AUC Total for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Non-compartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The AUC total was calculated as the sum of AUC0-96hr following the Day 1 dose and AUCinf following the Day 5 dose.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 0 | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 4 | 5 | 3 | 3
hr*ng/mL |  | 1.62 | 2.22 (1.05) | 2.59 (NA) — Not calculated when N = 2 | 10.8 (NA) — Not calculated when N = 2 | 35.6 (26.4) | 28.8 (16.4) | 25.5 (NA) — Not calculated when N = 2 | 51.1 (16.6) | 71.2 (18.9) | 126 (42.7) | 51.2 (6.39)

9. Secondary Outcome: Schedule A: Terminal Half-life (T1/2,z) of Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Non-compartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  Terminal half-life (t1/2,z) was calculated as t1/2,z = ln(2)/λz, where λz is the first-order terminal rate constant estimated via linear regression of the terminal log-linear phase.
Time Frame: Cycle 1 day 5 at predose and 1, 6, 12, 24, 48, 72, and 312 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 0 | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 4 | 5 | 3 | 4
hours |  | 16.3 | 35.1 (21.7) | 14.3 (NA) — Not calculated when N = 2 | 35.2 (NA) — Not calculated when N = 2 | 54.7 (20.5) | 55.8 (38.3) | 46.5 (NA) — Not calculated when N = 2 | 36.5 (13.3) | 41.7 (17.8) | 36.8 (22.4) | 40.6 (15.2)

10. Secondary Outcome: Schedule A: Clearance (CL) of Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Non-compartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  Clearance was calculated as Dose/λz*AUCinf.
Time Frame: Cycle 1 day 5 at predose and 1, 6, 12, 24, 48, 72, and 312 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab
Number analyzed (Participants) | 0 | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 4 | 5 | 3 | 4
mL/hr |  | 191 | 300 (66.2) | 963 (NA) — Not calculated when N = 2 | 742 (NA) — Not calculated when N = 2 | 584 (434) | 897 (718) | 1330 (NA) — Not calculated when N = 2 | 1420 (474) | 2070 (611) | 2210 (1030) | 1980 (459)

11. Secondary Outcome: Schedule B: Maximum Observed Concentration (Cmax) of Emerfetamab
Description: as for outcome 4
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 3
ng/mL | 4.07 | 4.71 (2.01)

12. Secondary Outcome: Schedule B: Time to Maximum Observed Concentration (Tmax) of Emerfetamab
Description: as for outcome 4
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 3
hours | 5.5 | 1.0 [1.0 to 6.3]

13. Secondary Outcome: Schedule B: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The area under the concentration-time curve from time 0 relative to the start of the IV infusion to the last quantifiable concentration was estimated using the linear trapezoidal method.
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 3
hr*ng/mL | 97.2 | 42.9 (20.4)

14. Secondary Outcome: Schedule B: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) for Emerfetamab
Description: Serum concentrations of emerfetamab were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (0.0015 ng/mL) were set to zero before data analysis.
  The area under the concentration-time curve from time 0 relative to the start of the IV infusion to infinity was estimated using the linear trapezoidal method.
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: Participants who received at least 1 dose of study drug, had at least 1 PK sample collected, with enough data for calculation of the PK parameter. No participants in Schedule B cohort 2 had data available for calculation of AUCinf.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 0
hr*ng/mL | 106 |

15. Secondary Outcome: Schedule B: Terminal Half-life (T1/2,z) of Emerfetamab
Description: as for outcome 4
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: Participants who received at least 1 dose of study drug, had at least 1 PK sample collected, with enough data for calculation of the PK parameter. No participants in Schedule B cohort 2 had data available for calculation of T1/2,z.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 0
hours | 30.5 |

16. Secondary Outcome: Schedule B: Clearance of Emerfetamab
Description: as for outcome 4
Time Frame: Cycle 1 day 14 at predose and 1, 6, 12, 24, 48, 72, 96, and 120 hours after the start of infusion.
Population: Participants who received at least 1 dose of study drug, had at least 1 PK sample collected, with enough data for calculation of the PK parameter. No participants in Schedule B cohort 2 had data available for calculation of clearance.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 0
mL/hr | 0.677 |

17. Secondary Outcome: Response Rate
Description: Disease response was based upon review of cytogenetics, bone marrow (BM) aspirates/biopsies, and peripheral blood count. Response rate is defined as the percentage of participants with a best overall response of complete remission (CR), CR with incomplete recovery (CRi) or morphologic leukemia-free state (MLFS) according to Revised International Working Group (IWG) response criteria, or CR with partial hematologic recovery (CRh*).
  CR: BM blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) > 1.0 x 10^9/L; platelet count > 100 x 10^9/L; independence of red cell transfusions.
  CRi: All CR criteria except residual neutropenia or thrombocytopenia. MLFS: BM blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required.
  CRh*: < 5% blasts in BM; no evidence of disease; partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl; no extramedullary disease.
Time Frame: Disease response was assessed on day 14 of every treatment cycle and at the end of study; median (min, max) duration was 1.22 (0.10, 5.98) months.
Population: All participants who received at least one dose of study drug.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3
percentage of participants | 0.0 [0.0 to 90.0] | 0.0 [0.0 to 90.0] | 0.0 [0.0 to 53.6] | 0.0 [0.0 to 53.6] | 0.0 [0.0 to 53.6] | 0.0 [0.0 to 53.6] | 0.0 [0.0 to 53.6] | 0.0 [0.0 to 53.6] | 25.0 [2.6 to 68.0] | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 43.8] | 0.0 [0.0 to 43.8] | 40.0 [11.2 to 75.3] | 0.0 [0.0 to 53.6]

18. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the interval from the date of the first disease assessment indicating an overall response to the first documented relapse or death due to any cause, whichever occurred first.
Time Frame: as for outcome 17
Population: All participants who received at least one dose of study drug with a best response of CR, CRi, MLFS, or CRh*
Measure: Median (Full Range); unit: days
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
days |  |  |  |  |  |  |  |  | 22 |  |  |  | 21 [1 to 41] |

19. Secondary Outcome: Time to Response
Description: Time to response is defined as the interval from the first administration of study drug to the first documentation of response. Time to response was evaluated only for participants who achieved a response.
Time Frame: as for outcome 17
Population: All participants who received at least one dose of study drug with a best response of CR, CRi, MLFS, or CRh*
Measure: Median (Full Range); unit: days
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
days |  |  |  |  |  |  |  |  | 42 |  |  |  | 22 [14 to 30] |

20. Secondary Outcome: Time to Progression
Description: Time to progression (event-free survival) is defined as the interval from first administration of study drug to the earliest of date of treatment failure, relapse for responders, or death due to any cause. For non-responders, the event date for treatment failure was assigned as the date of first administration of study drug.
Time Frame: as for outcome 17
Population: All participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 4 | 5 | 3
days | 1 | 1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 63] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 11] | 1 [1 to 70] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment until end of study; median (min, max) time on study was 1.31 (0.20, 5.98) months. Adverse events are reported from first dose of study drug until the end of study; median (min, max) duration was 1.22 (0.10, 5.98) months.
Arm/Group | Schedule A Cohort 1: 0.05 µg Emerfetamab | Schedule A Cohort 2: 0.15 µg Emerfetamab | Schedule A Cohort 3: 0.45 µg Emerfetamab | Schedule A Cohort 4: 1.5 µg Emerfetamab | Schedule A Cohort 5: 4.5 µg Emerfetamab | Schedule A Cohort 6: 7 µg Emerfetamab | Schedule A Cohort 7: 9 µg Emerfetamab | Schedule A Cohort 8: 18 µg Emerfetamab | Schedule A Cohort 9: 36 µg Emerfetamab | Schedule A Cohort 10: 72 µg Emerfetamab | Schedule A Cohort 11: 110 µg Emerfetamab | Schedule A Cohort 12: 36/72 µg Emerfetamab | Schedule B Cohort 1: 72 µg Emerfetamab | Schedule B Cohort 2: 110 µg Emerfetamab
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/4 | 0/6 | 0/4 | 1/4 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/3 | 1/3 | 2/3 | 1/3 | 2/3 | 3/3 | 2/4 | 5/6 | 3/4 | 4/4 | 1/5 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 4/4 | 4/4 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A Cohort 1: 0.05 µg Emerfetamab (N=1) | Schedule A Cohort 2: 0.15 µg Emerfetamab (N=1) | Schedule A Cohort 3: 0.45 µg Emerfetamab (N=3) | Schedule A Cohort 4: 1.5 µg Emerfetamab (N=3) | Schedule A Cohort 5: 4.5 µg Emerfetamab (N=3) | Schedule A Cohort 6: 7 µg Emerfetamab (N=3) | Schedule A Cohort 7: 9 µg Emerfetamab (N=3) | Schedule A Cohort 8: 18 µg Emerfetamab (N=3) | Schedule A Cohort 9: 36 µg Emerfetamab (N=4) | Schedule A Cohort 10: 72 µg Emerfetamab (N=6) | Schedule A Cohort 11: 110 µg Emerfetamab (N=4) | Schedule A Cohort 12: 36/72 µg Emerfetamab (N=4) | Schedule B Cohort 1: 72 µg Emerfetamab (N=5) | Schedule B Cohort 2: 110 µg Emerfetamab (N=3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 2 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A Cohort 1: 0.05 µg Emerfetamab (N=1) | Schedule A Cohort 2: 0.15 µg Emerfetamab (N=1) | Schedule A Cohort 3: 0.45 µg Emerfetamab (N=3) | Schedule A Cohort 4: 1.5 µg Emerfetamab (N=3) | Schedule A Cohort 5: 4.5 µg Emerfetamab (N=3) | Schedule A Cohort 6: 7 µg Emerfetamab (N=3) | Schedule A Cohort 7: 9 µg Emerfetamab (N=3) | Schedule A Cohort 8: 18 µg Emerfetamab (N=3) | Schedule A Cohort 9: 36 µg Emerfetamab (N=4) | Schedule A Cohort 10: 72 µg Emerfetamab (N=6) | Schedule A Cohort 11: 110 µg Emerfetamab (N=4) | Schedule A Cohort 12: 36/72 µg Emerfetamab (N=4) | Schedule B Cohort 1: 72 µg Emerfetamab (N=5) | Schedule B Cohort 2: 110 µg Emerfetamab (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intravascular haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 2 | 2 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 5 | 3 | 2 | 5 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Genital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time shortened (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 2 | 3 | 2 | 1 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 4 | 1 | 2 | 2
Blast cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03224819/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03224819/SAP_001.pdf